CLINICAL TRIAL: NCT07266259
Title: Effects of Levocarnitine and Myoinositol in Comparison to Myoinositol Alone on Hormonal and Insulin Resistance Parameters in Subfertile Women With Insulin Resistant Polycystic Ovary Syndrome
Brief Title: Effect of Levocarnitine Plus Myoinositol Versus Myoinositol Alone on Hormonal and Insulin Resistance in PCOS Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mst.Sumyara Khatun (Other)
Responsible Party: Sponsor-Investigator, Mst.Sumyara Khatun, Medical Officer, Bangladesh Medical University
Organization: Bangladesh Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5722
Record Dates: First submitted 2025-09-21; First posted 2025-12-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: levocarnitine myoinositol; insulin resistance hormonal parameters; polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm:( Levocarnitine and myoinositol) (Experimental): Participants will receive levocarnitine 330mg and myoinositol 750mg twice daily for 3 months
  Interventions: Combination Product: Levo-Carnitine
- Active Comparator (Myoinositol) (Active Comparator): Participants will receive myoinositol 750mg twice daily for 3 months
  Interventions: Dietary Supplement: Myoinositol

INTERVENTIONS:
Dietary Supplement: Myoinositol — Myoinositol 750mg twice daily for 3 months
  Arms: Active Comparator (Myoinositol)
Combination Product: Levo-Carnitine — Levocarnitine 330 mg and Myoinositol 750 mg twice daily for 3 months
  Other Names: Myoinositol
  Arms: Experimental arm:( Levocarnitine and myoinositol)

SUMMARY:
The goal of this clinical trial is to learn if combination of levocarnitine and myoinositol works better than myoinositol alone on insulin resistance and hormonal parameters in subfertile women with insulin resistant polycystic ovary syndrome . It will also learn about the safety of drug levocarnitine and myoinositol. The main questions it aims to answer are:

Does combined action of levocarnitine and myoinositol improve insulin resistance and hormonal parameters in comparison to myoinositol alone in subfertile women with insulin resistant polycystic ovary syndrome ? What medical problems do participants have when taking drug levocarnitine and myoinositol? Researchers will compare the drug combination of levocarnitine and myoinositol to myoinositol alone to see if combination therapy works better?

Participants will:

Take drug levocarnitine and myoinositol or a myoinositol alone twice daily for 3 months Visit the clinic once after 3 months for checkups and tests Keep a diary of their symptoms and the number of times.

DETAILED DESCRIPTION:
After obtaining approval of the Institutional Review Board, this randomized controlled trial will be conducted in the department of Reproductive Endocrinology & Infertility,,Bangladesh Medical University (BMU), Shahbag,Dhaka. A total number of 72 subfertile women with insulin resistance polycystic ovary syndrome, after fulfilling the inclusion and exclusion criteria will be approached for informed written consent after discussing the purpose and procedure of the study. This patient will be collected from REI outdoor department of Reproductive Endocrinology & Infertility, BMU.Every patient will be asked to come fasting on a particular day, time, and place. Related history will be taken and physical examination (height, weight, waist circumference, hip circumference, acne, hirsutism, acanthosis nigricans) will be done and all data will be documented in a pretested semi-structured questionnaire.

After adequate preparation and precaution, about 04 ml of venous blood will be drawn from each participant after 8-12 hours of fasting.

About4 ml of whole blood collected during fasting, 2 ml will be kept in a fluorinated tube for measuring fasting blood glucose (FBG), and 2 ml of blood for serum collection, will be kept standing for 15 minutes to allow clotting before centrifugation. After centrifugation, the serum will be separated and kept in microcentrifuge tubes. After proper labeling, the fluorinated tube and adequate serum will be tested for fasting blood sugar andserum fasting insulin on the same collection day in department of biochemistry and molecular biology,BMU.Fasting blood glucose by glucose oxidase method,fasting insulin by chemiluminescent technology by atellicaIM IRI assay in BMU. Then HOMA-IR will be calculated.If HOMA-IR index >2.6 ,then patient will be asked to come on their second day of menstruation.After adequate preparation and precaution, about 4 ml of venous blood will be drawn from each participant,will be kept standing for 15 minutes to allow clotting before centrifugation. After centrifugation, the serum will be separated and kept in microcentrifuge tubes. After proper labeling, adequate serum will be tested for serum follicle stimulating hormone(FSH),serum luteinizing hormone(LH) by chemiluminescence immunoassay(ADVIA Centaur XPT Immunoassay) and serum free testosterone level by chemiluminescence (MAGLUMI X8) on the same collection day in microbiology & immunology department of BMU.

Detailed socio-demographic data, history,examination findings and investigations will be recorded in a predesigned data sheet.

Eligible women who will give their informed consent will be randomized into two groups. Allocation concealment will be done by serially numbered sealed envelopes. Each envelope will be labeled with a serial number and will have a card noting the intervention type. Allocation will never be changed after opening the sealed envelopes.

The experimental group will be treated with levocarnitine 330mg and myoinositol 750mg twice daily for 3 months.The comparator group will be treated with myoinositol 750 mg twice daily alone for 3 months.Then monthly over phone follow-up will be given about the patient's compliance. Any adverse events or side effects related to supplementation will be recorded and managed accordingly.

They will also be informed not to take other medications except after consulting with us.

After 3 months of intervention patients will come at Reproductive Endocrinology Infertility department on their second day(D2) of menstruation with 8-12 hours fasting. Then I will check strip of drug whether patient had taken the drug properly or not. Fasting blood sugar,fasting insulin,serum FSH,LH,free testosterone will be done by the same procedure.

Then data will be collected from the patients on using interviews, observation, clinical examination, investigations. The cumulative data will be subjected to analysis. All the clinical, biochemical and hormonal information will be documented in a pretested,semi structured clinical case record form.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-40 years old.
* Diagnosed cases of PCOS patients(both old & new cases) according to International evidence-based guideline criteria 2023
* Primary or secondary subfertility.
* Insulin resistance (HOMA-IR >2.6)

Exclusion Criteria:

* Hypothyroidism
* Diabetes mellitus
* Hormonal (Myo-inositol,D-chiro-inositol) or insulin sensitizing drugs like Metformin,Pioglitazone etc. treatment in the last three months
* Known hypersensitivity to Myo-inositol and Levo-carnitine
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 72 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in homeostatic model assessment of Insulin Resistance (HOMA-IR) | Baseline to 12 weeks after treatment
  HOMA-IR will be calculated as (fasting insulin(micro IU/mL*fasting glucose(mmol/L)/22.5

SECONDARY OUTCOMES:
Change in serum LH level | Baseline and after 12 weeks of treatment
  Serum LH level will be measured on day 2 of the menstrual cycle by Chemiluminescence immunoassay [ADVIA Centaur XPT ImmunoassaySystem].D2-D5 Serum LH-5-20IU/L.
Change in serum FSH level | baseline and 12 weeks after treatment
  Serum FSH level will be measured on day 2of the menstrual cycle by Chemiluminescence immunoassay [ADVIA Centaur XPTImmunoassay System].(D2-D5) Serum FSH-5-20IU/L
Change in LH:FSH ratio | baseline and 12 weeks after treatment
  The LH/FSH ratio will be calculated by dividing serum LH (mIU/mL) by FSH mIU/mL).
Change in serum free testosterone | baseline and 12 weeks after treatment
  Free testosterone will bemeasured on menstrual day 2 by Chemiluminescence immunoassay [MAGLUMI X8, Germany]. Normal value for a female is 0.7 to 3.6 pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jemine Banu, MS, Study Director — Bangladesh Medical University
Locations (1):
- Bangladesh Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Genazzani AD, Battipaglia C, Foschi M, Semprini E, Aio C, Spelta E, Kostrzak A, Rusce ML, Szeliga A, Meczekalski B. Improved insulin sensitivity and reproductive profile in overweight/obese PCOS patients undergoing integrative treatment with carnitines, L-arginine, L-cysteine and myo-inositol. Gynecol Endocrinol. 2025 Dec;41(1):2458710. doi: 10.1080/09513590.2025.2458710. Epub 2025 Jan 28. PMID 39874141
- [Background] Agarwal A, Sengupta P, Durairajanayagam D. Role of L-carnitine in female infertility. Reprod Biol Endocrinol. 2018 Jan 26;16(1):5. doi: 10.1186/s12958-018-0323-4. PMID 29373970